CLINICAL TRIAL: NCT06603298
Title: Evaluation of the Efficacy and Safety of Endoscopic Dilatation Combined With Biological Therapy Therapy for the Treatment of Intestinal Stenosis in Patients With Crohn's Disease
Brief Title: Evaluation of the Efficacy and Safety of Endoscopic Dilatation and Biological Therapy in Intestinal Stenosis Due to CD
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ENDO_BIO- CROHN- ID 6815
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-09

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical therapy alone: It includes patients with Crohn's disease who were only treated with biological therapy for clinically significant intestinal stenosis. These patients underwent drug treatment without any endoscopic procedure.
- Medical therapy + endoscopic dilatation: It includes patients who received both endoscopic dilatation (ED) with a balloon and biological therapy. This cohort underwent combined treatment for intestinal stenosis, integrating mechanical and pharmacological intervention.

SUMMARY:
All patients with Crohn's disease, already undergoing biological therapy for the treatment of clinically significant intestinal stenosis and/or already undergoing endoscopic balloon dilatation during the period January 2016 - June 2024 will be enrolled.

DETAILED DESCRIPTION:
All patients meeting all inclusion criteria and no exclusion criteria will be offered participation in the study upon presentation of the information form and signing of the informed consent for participation in the study. Each patient will be assigned a progressive identification number (ID).

All clinical data will be recorded for all patients:

* Demographic data (age, sex, smoking habits)
* Montreal classification;
* Duration of disease;
* History of previous surgery;
* Past and current drug therapy.

All available data on stenosis characteristics will be recorded:

* Localisation (ileal, ileo-caecal, colic, anastomotic);
* Extent (mm);
* Evidence of concurrent endoscopic disease activity locally

All data related to the endoscopic procedure will also be recorded:

* Size of device used;
* Maximum dilatation achieved (mm);
* Technical success, assessed by endoscopic clearance of the stenosis after the dilation procedure;
* Consensual local steroid injection;
* Possible multiple endoscopic dilation sessions;

The occurrence of episodes of intestinal sub-occlusion or occlusion will be recorded, the introduction of steroid therapy and the need for surgery. Where available radiological and endoscopic re-evaluation data will be recorded.

Any changes in treatment and any adverse events, defined as any adverse event, will also be recorded. as any adverse event without a necessary causal relationship with the endoscopic procedure and the concomitant ongoing biological therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Confirmed diagnosis of Crohn's disease;
* Radiological or endoscopic evidence of Crohn's disease complicated by clinically significant intestinal stenosis treated by endoscopic balloon dilatation.
* Minimum 12-month clinical follow-up at this hospital;
* Ability to express and give informed consent for participation in the study and to adhere to the timetable of scheduled visits.

Exclusion Criteria:

* Age <18 years;
* Patients with pouch or terminal ileostomy;
* Any clinical condition that, in the opinion of the investigators, may contraindicate enrolment in the study;
* Unstable personality or inability to adhere to protocol procedures;
* Inability to express and give informed consent for study participation and to adhere to the participation in the study and to adhere to the timing of the planned visits.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with Crohn's disease
Sampling Method: Probability Sample
Enrollment: 182 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-10-17 (Estimated); Study Completion 2025-10-17 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with transitable colonoscopy at 12 months assessed by endoscopic and radiological documentation | 12 months
  Measurement of the percentage of patients with Crohn's disease and intestinal stenosis who obtain a transitable colonoscopy after 12 months of follow-up, comparing two interventions: single biological therapy vs. endoscopic dilatation combined with biological therapy. Transitability of the colonoscopy will be determined by the ability of the colonoscope to completely pass through the stenosis as documented in the endoscopic and/or radiological reports. Data will be aggregated as the proportion of patients with transitable colonoscopy in the total number of patients in each treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Scaldaferri, PI, Principal Investigator — Fondazione Policlinico Gemelli, Rome
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC CEMAD, Roma, Italy